CLINICAL TRIAL: NCT01117610
Title: A Preemptive Epidural Ropivacaine for Postoperative Pain Relief in Degenerative Lumbar Spine Surgery: A Prospective Randomized Study
Brief Title: A Preemptive Epidural Ropivacaine for Postoperative Pain Relief in Degenerative Lumbar Spine Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Kwang-Sup Song, Chung-Ang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChungAngUH
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Postoperative Pain
Keywords: pain; preemptive; postoperative; epidural injection; laminectomy
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ropivacaine; Injections, Epidural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- epidural injection (group I) (Active Comparator): patients in Group I will receive epidural injection of 0.1% ropivacaine 10 ml before skin incision.
  Interventions: Drug: Ropivacaine (epidural injection)
- epidural injection group (group C) (Placebo Comparator): control group will receive no medication preoperatively and during operation
  Interventions: Drug: Placebo (one of medication)

INTERVENTIONS:
Drug: Placebo (one of medication) — patients in Group C will receive none of medication preoperatively and intraoperatively
  Other Names: patient in group C will receive none of medication
  Arms: epidural injection group (group C)
Drug: Ropivacaine (epidural injection) — patient in group I will receive epidural injection of 0.1% ropivacaine 10ml before skin incision.
  Other Names: epidural injection
  Arms: epidural injection (group I)

SUMMARY:
This prospective randomized study aims to evaluate the effectiveness of epidural injection of ropivacaine on the relief of pain in patients undergoing laminectomy.

Total 60 patients will be randomized into one of two groups (groupC or groupI) based on Excel number generation.

Patients in group C will receive no medication intraoperatively, and patients in group I will receive epidural injection of 0.1% ropivacaine 10ml before skin incision.

Visual analogue scale pain scores, fentanyl consumption and the frequency at which patients pushed the button (FPB) of a patient-controlled analgesia system will be recorded at 4,12,24,48 hour postoperatively.

DETAILED DESCRIPTION:
Patients in group I will receive 0.1% ropivacaine 10 ml before skin incision under guide of C-arm.

ELIGIBILITY:
Inclusion Criteria:

* laminectomy

Exclusion Criteria:

* r/o infection
* reoperation
* mental change
* allergy to local anesthetics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale 4hour | post op 4hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 4hour.

SECONDARY OUTCOMES:
visual analogue scale 24hour | Post Op 24 hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 24hour.
visual analogue scale 12 hour | Post op 12 hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 12 hour.
Visual analogue scale 48hour | Post Op 48hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 48 hour.
Opioid consumption 4hour | Post Op 4hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid fom immediately after operation to post op 4hour will be measured.
Opioid consumption 24hour | Post op 24 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid from 12 hour to post op 24 hour will be measured.
Opioid consumption 12 hour | Post Op 12 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid from post op 4hour to post op 12 hour will be measured.
Opioid consumption 48hour | Post Op 48 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid from post op 24 hour to post op 48 hour will be measured
FPB 4 hour | Post Op 4 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 4 hour will be measured.
FPB 12 hour | post op 12 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And frequency of patient to push the button of the PCA machine (FPB) from post op 4 hour to post op 12 hour will be measured.
FPB 24 hour | Post Op 24 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And frequency of patient to push the button of the PCA machine (FPB) fom post op 12 hour to post op 24 hour will be measured.
FPB 48 hour | Post Op 48 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And frequency of patient to push the button of the PCA machine (FPB) fom post op 24 hour to post op 48 hour will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-Sup Song, M.D. & Ph.D., Study Director — ChungAng University; Hyun Kang, M.D. & Ph.D., Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- ChungAng University, Seoul, South Korea

REFERENCES:
- [Derived] Kang H, Jung HJ, Lee JS, Yang JJ, Shin HY, Song KS. Early postoperative analgesic effects of a single epidural injection of ropivacaine administered preoperatively in posterior lumbar interbody spinal arthrodesis: a pilot randomized controlled trial. J Bone Joint Surg Am. 2013 Mar 6;95(5):393-9. doi: 10.2106/JBJS.K.01729. PMID 23467861